CLINICAL TRIAL: NCT06822491
Title: Early Magnetic Resonance Imaging Response of the Dominant Intraprostatic Lesion After Online Adaptive Stereotactic Body Radiotherapy for Localized Prostate Cancer and Correlation With Prostate Specific Antigen Response (PRODART)
Brief Title: Early Magnetic Resonance Imaging Response of the Dominant Intraprostatic Lesion After Online Adaptive Stereotactic Body Radiotherapy for Localized Prostate Cancer and Correlation With Prostate Specific Antigen Response
Acronym: PRODART
Status: Active, not recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: RAO-24-005
Record Dates: First submitted 2025-02-06; First posted 2025-02-12 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Prostate Carcinoma; Localized Prostate Adenocarcinoma; Stereotactic Body Radiotherapy; Stereotactic Radiotherapy; Magnetic Resonance Imaging; Multiparametric MRI
Keywords: DIL; Dominant intraprostatic lesion
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this phase II study is to determine the early multiparametric magnetic resonance imaging response of the dominant intraprostatic lesion and correlate these findings with prostate specific antigen response in patients with intermediate to (very) high risk localized prostate cancer treated with online adaptive stereotactic radiotherapy without intraprostatic fiducial markers.

DETAILED DESCRIPTION:
Background: Stereotactic body radiotherapy (SBRT) is an established standard of care treatment for localized prostate cancer. Recent pathological studies suggest the presence of a dominant intraprostatic lesion (DIL) within the prostate, which serve as a central driver of tumor aggressiveness and recurrence after treatment. Prostate-specific antigen (PSA) monitoring is the cornerstone of follow-up, though time to PSA nadir after SBRT can extend to 3 years.

Methods: This phase II observational study aims to evaluate the correlation between PSA response and early multiparametric magnetic resonance imaging (mpMRI) changes of the DIL(s) at 6- or 9-months following online adaptive SBRT for intermediate to (very) high risk localized prostate cancer. The primary outcome is the achievement of local control as assessed by mpMRI at 6 months post-SBRT or, if necessary, at 9 months post-SBRT (in case of image non complete response at 6 months). A complete imaging response is defined as the disappearance of all morphological and functional mpMRI changes of PIRADS (Prostate Imaging Reporting and Data System) ≥3 lesion(s) correlating with Gleason ≥7a pathology. No confirmatory biopsies will be conducted. The required sample size for this study will be 28 patients, assuming a complete response rate of 80% at 6 months, targeting an acceptable margin of error with 95% confidence, and a margin of error of 15%.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed localized prostate cancer who are planned for CT- or MRI-adaptive SBRT for prostate cancer;
* Presence of PIRADS ≥3 lesion(s) in a mpMRI correlating with Gleason ≥7 score at diagnosis;
* Intermediate to (very) high risk localized prostate cancer (≤ cT3b and cN0);
* ECOG performance status of 0-2;
* Age ≥ 18 years;
* PSMA PET ≤3 months is compulsory for high-risk prostate cancer (as part of clinical routine);
* Written informed consent.
* Willingness and ability to comply with schedule

Exclusion Criteria:

* Previous (≤10 years) local therapy of the prostate including transurethral resection of the prostate (TURP),
* Contraindication for MRI;
* Previous (≤10 years) radiotherapy in the pelvis;
* Lymph node metastases or distant metastases (i.e. no localized prostate cancer);
* Participation in a clinical trial which might influence the results of this project;
* Claustrophobic anxiety;
* Uncontrolled intercurrent illness;
* Relation to investigator (family or professional)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to our tertiary referral centre for prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Multiparametric magnetic resonance imaging local control of the dominant intraprostatic lesion | 6 months after SBRT. In cases with image non-complete response at 6 months, 3 months later (in total 9 months after SBRT) an additional mpMRI will be performed.
  To study multiparametric magnetic resonance imaging (mpMRI) local control of Prostate Imaging Reporting and Data System (PIRADS) ≥3 lesion(s) after SBRT. An image complete response is defined as disappearance of all morphological and functional PIRADS ≥3 lesion(s) correlating with Gleason ≥7a pathology in mpMRI.
Correlation of early prostate-specific antigen response with early multiparametric magnetic resonance imaging changes | 6 months after SBRT. In cases with image non-complete response at 6 months, 3 months later (in total 9 months after SBRT) an additional mpMRI will be performed.
  To correlate early prostate-specific antigen response with early multiparametric magnetic resonance imaging changes of the PIRADS ≥3 lesion(s) correlating with Gleason ≥7a pathology

SECONDARY OUTCOMES:
Correlation of late prostate-specific antigen response with early multiparametric magnetic resonance imaging changes | Yearly (up to 5 years post SBRT)
  To correlate late prostate-specific antigen response with early multiparametric magnetic resonance imaging changes of the PIRADS ≥3 lesion(s) correlating with Gleason ≥7a pathology
Correlation of genitourinary and gastrointestinal toxicity with early multiparametric magnetic resonance imaging changes | 6 months after SBRT. In cases with image non-complete response at 6 months, 3 months later (in total 9 months after SBRT) an additional mpMRI will be performed.
  Correlating genitourinary and/or gastrointestinal toxicity (according to common terminology criteria for adverse events [CTCAE] version 5.0) with structural and/or functional changes of the prostate and/or surrounding organs on early multiparametric magnetic resonance imaging
Correlation of prostate quality of life with early multiparametric magnetic resonance imaging changes | 6 months after SBRT. In cases with image non-complete response at 6 months, 3 months later (in total 9 months after SBRT) an additional mpMRI will be performed.
  Quality of life (according to EPIC-26) and relation to early structural and/or functional changes of the prostate and/or surrounding organs on multiparametric magnetic resonance imaging
To evaluate prostate volume change during and after adaptive prostate SBRT and to correlate to treatment toxicity. | Intra-treatment (within 1 week before the last fraction of SBRT) and 6 months after SBRT. In cases with image non-complete response at 6 months, 3 months later (in total 9 months after SBRT) an additional mpMRI will be performed.
  To evaluate prostate volume change intra-treatment and after adaptive prostate SBRT and to correlate to treatment toxicity.
Exploratory image analysis | 6 months after SBRT. In cases with image non-complete response at 6 months, 3 months later (in total 9 months after SBRT) an additional mpMRI will be performed.
  Quantitative imaging features will be used to predict outcome and side effects on the different images.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Guckenberger, Prof. Dr. med., Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this trial after de-identification. Other documents may be shared include the study protocol.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months after article publication.
Access Criteria: Proposals to access study data should send request to matthias.guckenberger@usz.ch. To gain access, data requesters must sign data access agreement.